CLINICAL TRIAL: NCT00812318
Title: A Single Dose, Randomized Study to Assess the Relative Bioavailability of Two Formulations and Food Effect on GSK1265744 in Healthy Male and Female Subjects
Brief Title: Healthy Volunteer Study To Assess The Bioavailability of GSK1265744 When Administered Orally Either When Fasted or Following a Meal.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: Shionogi (Industry); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ITZ111682
Record Dates: First submitted 2008-09-05; First posted 2008-12-22 (Estimated); Last update posted 2012-04-02 (Estimated); Status verified 2012-03

CONDITIONS: HIV Infection; Infection, Human Immunodeficiency Virus
Keywords: HIV infected subjects; Healthy volunteer; GSK1265744.
MeSH Terms: conditions — HIV Infections; Infections; Acquired Immunodeficiency Syndrome | interventions — cabotegravir; Solutions; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment A (Experimental): GSK1265744 10mg oral solution
  Interventions: Drug: GSK1265744 10 mg oral solution
- Treatment B (Experimental): GSK1265744 5mg tablet, fasted
  Interventions: Drug: GSK1265744 5 mg tablet
- Treatment C (Experimental): GSK1265744 5mg tablet, fed
  Interventions: Drug: GSK1265744 5 mg tablet

INTERVENTIONS:
Drug: GSK1265744 10 mg oral solution — GSK1265744
  Other Names: GSK1265744
  Arms: Treatment A
Drug: GSK1265744 5 mg tablet — GSK1265744 5mg tablet, fasted
  Other Names: GSK1265744
  Arms: Treatment B
Drug: GSK1265744 5 mg tablet — GSK1265744 5mg tablet, fed
  Other Names: GSK1265744
  Arms: Treatment C

SUMMARY:
To evaluate the single dose relative bioavailability of GSK1265744 10mg administered in either oral solution fasted, two 5mg tablets fasted, or two 5mg tablets following a moderate meal.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible physician, based on a medical evaluation including medical history, physical examination, laboratory tests and 12-lead ECG. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Male or female between 18 and 55 years of age.
* A female subject is eligible to participate if she is of non-childbearing potential (i.e., physiologically incapable of becoming pregnant) including any female who:

  * Is pre-menopausal with a documented bilateral tubal ligation, bilateral oophorectomy (removal of the ovaries) or hysterectomy, or
  * Is post-menopausal defined as 12 months of spontaneous amenorrhea. A follicle stimulating hormone (FSH) level will be performed to confirm a post-menopausal status. For this study, FSH levels > 40 mlU/ml is confirmatory.
* A male is eligible to enter and participate in the study if he is surgically sterile OR if he either agrees to abstain from sexual intercourse with a female partner or agrees to use a condom/spermicide, in addition to having his female partner use another form of contraception as outlined in Section 7.1.
* Body weight >= 50 kg (110 lbs.) for men and >= 45 kg (99 lbs) for women and body mass index (BMI) within the range 18.5-31.0 kg/m2 (inclusive).
* A signed and dated written informed consent is obtained from the subject or the subject's legal representative prior to screening.
* Subject must be capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

* As a result of the medical interview, physical examination, or screening investigations, the Investigator considers the subject unfit for the study.
* Has a positive pre-study Hepatitis B surface antigen; positive hepatitis C (HCV) antibody or detectable HCV ribonucleic acid (RNA); or positive HIV-1 antibody result.
* Has a history of regular alcohol consumption averaging >7 drinks/week for women or >14 drinks/week for men within 6 months of the screening visit.

Note: 1 drink is equivalent to 12 g alcohol = 5 ounces (150 ml) of wine or 12 ounces (360 ml) of beer or 1.5 ounces (45 ml) of 80 proof distilled spirits.

* Unwilling to abstain from alcohol for 48 hours prior to the start of dosing until collection of the final pharmacokinetic sample during each treatment period.
* Unwilling to refrain from the use of illicit drugs and adhere to other protocol-stated restrictions while participating in the study.
* The subject has received an investigational drug or participated in any other research trial within 30 days or 5 half-lives, or twice the duration of the biological effect of any drug (whichever is longer) prior to the first dose of current study medication.
* Participation in the study would result in donation of blood in excess of 500 mL within a 56 day period.

Note: This does not include plasma donation.

- History or presence of allergy or intolerance to the study drug or its components or drugs of its class, or a history of drug or other allergy that, in the opinion of the physician responsible, contraindicates their participation. In addition, if heparin is used during PK sampling, subjects with a history of sensitivity to heparin or heparin-induced thrombocytopenia should not be enrolled.

Note: "Study" or "investigational" drugs include GSK1265744 or placebo.

* Subjects with a pre-existing condition interfering with normal gastrointestinal anatomy or motility, hepatic and/or renal function, that could interfere with the absorption, metabolism, and/or excretion of the study drugs. Subjects with a history of cholecystectomy should be excluded.
* Exclusion criteria for screening ECG per protocol
* The subject's systolic blood pressure is outside the range of 90-140mmHg, or diastolic blood pressure is outside the range of 45-90mmHg or heart rate is outside the range of 50-100bpm for female subjects or 45-100 bpm for male subjects.
* Has a history of regular use of tobacco- or nicotine-containing products within 3 months of the screening visit.
* The subject has a positive pre-study drug and/or alcohol screen.
* Use of prescription or non-prescription drugs, including antacids, vitamins, herbal and dietary supplements (including St John's Wort and iron supplements) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and sponsor the medication will not interfere with the study procedures or compromise subject safety

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2008-06; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Composite of pharmacokinetic parameters | 6 days
  Plasma GSK1265744 Area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time [AUC(0-infinity)], Area under the concentration-time curve over the dosing interval [AUC(0-t)], and Maximum observed concentration (Cmax).

SECONDARY OUTCOMES:
Safety and tolerability parameters, including the collection adverse events | 6 days
Composite of pharmacokinetic parameters | 6 days
  Plasma GSK1265744 Terminal phase half-life (t½), Lag time before observation of drug concentrations in sampled matrix (tlag), Time of occurrence of Cmax (tmax), and Apparent clearance following oral dosing (CL/F).
Safety and tolerability parameters including the change from baseline in clinical laboratory assessments | 6 days
  Clinical chemistry, hematology and urinalysis compared to baseline values
Safety and tolerability parameters including the collection of concurrent medication | 6 days
Safety and tolerability parameters including the change from baseline in electrocardiogram values (ECG). | 6 days
Safety and tolerability parameters including change from baseline in vital sign measurements | 6 days
  blood pressure and heart rate

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Buffalo, New York, United States